CLINICAL TRIAL: NCT02642133
Title: Breastfeeding Improvement Following Tongue-tie and Lip-tie Release: A Prospective Cohort Study
Brief Title: Breastfeeding Improvement Following Tongue-tie and Lip-tie Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Oregon Clinic (Other)
Responsible Party: Principal Investigator, Bobak Ghaheri, MD, Otolaryngologist, The Oregon Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOC ENT
Record Dates: First submitted 2015-12-22; First posted 2015-12-30 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Ankyloglossia; Breastfeeding
MeSH Terms: conditions — Ankyloglossia; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Other): All patients were in the same arm - this is a cohort study where the group serves as their own control. Patients who did not undergo the procedure were not included in this outcomes study.
  Interventions: Procedure: Lingual Frenotomy and/or maxillary labial frenectomy

INTERVENTIONS:
Procedure: Lingual Frenotomy and/or maxillary labial frenectomy — The procedure is performed with a 1064nm InGaAsP semiconductor diode laser which is a soft tissue laser with variable pulsed wave and wattage settings. The procedure was performed at 0.7-0.8 pulsed watts, 200 microseconds on and 100 microseconds off (actual wattage: 0.47 to 0.53 W) using a 300 micron laser fiber. The tongue is elevated using a grooved director while the laser tip is applied to the frenulum. If present, the anterior frenulum is divided until the submucosal portion of the tie is identified (this is the posterior tongue-tie). A small window in the central mucosa is made and the lateral mucosal walls of the posterior tongue-tie are released, taking care to not disturb the fascia of the underlying genioglossus muscle.

SUMMARY:
This study is an observational study to determine outcomes of surgical release of tongue-tie and lip-tie in babies who are experiencing difficulty with breastfeeding.

DETAILED DESCRIPTION:
Breastfeeding rates in the United States initiate at around 80%, but many mothers are unable to effectively breastfeeding because of problems with latch and suction generation. Previous studies have demonstrated how nipple pain is directly linked to ankyloglossia, but most of these studies are done with poor methodology.

Clinically, tongue-tie and lip-tie have correlate with numerous other symptoms besides nipple pain. These babies tend to be inefficient nursers, which can affect weight gain. Abnormal intake of air because of the poor latch/seal can lead to reflux symptoms. Finally, there is a significant psychological toll on mothers who want to breastfeed but cannot do so.

This study aims to prospectively analyze these outcomes by using validated tools.

ELIGIBILITY:
Inclusion Criteria:

* Healthy babies who are breastfeeding 0-12 weeks of age

Exclusion Criteria:

* Serious comorbid conditions (heart, lung, brain)
* Prior maternal breast surgery
* Insufficient glandular tissue
* Previous tongue/lip surgery
* Twins/Triplets

Ages: 1 Day to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 237 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Nipple Pain | 1 week
  Using a visual analog scale, nipple pain is evaluated.
Reflux/GERD | 1 week
  Using a validated questionnaire (i-GERQ-R)
Breastfeeding efficiency | 1 week
  Volume of breastmilk ingested in a specific time frame calculated (mL/min)
Breastfeeding self-efficacy | 1 week
  Uses the BSES-SF validated questionnaire

SECONDARY OUTCOMES:
Nipple Pain | 1 month
  Using a visual analog scale, nipple pain is evaluated.
Reflux/GERD | 1 month
  Using a validated questionnaire (i-GERQ-R)
Breastfeeding self-efficacy | 1 month
  Uses the BSES-SF validated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Bobak A Ghaheri, MD, Principal Investigator — The Oregon Clinic

REFERENCES:
- [Background] O'Callahan C, Macary S, Clemente S. The effects of office-based frenotomy for anterior and posterior ankyloglossia on breastfeeding. Int J Pediatr Otorhinolaryngol. 2013 May;77(5):827-32. doi: 10.1016/j.ijporl.2013.02.022. Epub 2013 Mar 22. PMID 23523198
- [Background] Geddes DT, Langton DB, Gollow I, Jacobs LA, Hartmann PE, Simmer K. Frenulotomy for breastfeeding infants with ankyloglossia: effect on milk removal and sucking mechanism as imaged by ultrasound. Pediatrics. 2008 Jul;122(1):e188-94. doi: 10.1542/peds.2007-2553. Epub 2008 Jun 23. PMID 18573859
- [Background] Pransky SM, Lago D, Hong P. Breastfeeding difficulties and oral cavity anomalies: The influence of posterior ankyloglossia and upper-lip ties. Int J Pediatr Otorhinolaryngol. 2015 Oct;79(10):1714-7. doi: 10.1016/j.ijporl.2015.07.033. Epub 2015 Jul 31. PMID 26255605
- [Derived] Ghaheri BA, Cole M, Fausel SC, Chuop M, Mace JC. Breastfeeding improvement following tongue-tie and lip-tie release: A prospective cohort study. Laryngoscope. 2017 May;127(5):1217-1223. doi: 10.1002/lary.26306. Epub 2016 Sep 19. PMID 27641715